CLINICAL TRIAL: NCT04160156
Title: Clinical Use of the Long-term Implantable Sensor Improves Glycated Hemoglobin and Time in Range in Patients With Type 1 Diabetes
Brief Title: Long-term, Implantable Sensor Improves Health Outcomes in Patients With T1D
Status: Completed | Type: Observational
Sponsor: University Magna Graecia (Other)
Responsible Party: Principal Investigator, Concetta Irace, Professor, University Magna Graecia
Other Study IDs: Long term implantable sensor
Record Dates: First submitted 2019-11-07; First posted 2019-11-12 (Actual); Last update posted 2019-11-12 (Actual); Status verified 2019-11

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Continuous glucose monitoring; sensor; glycated hemoglobin; Time in range
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Type 1 diabetes: Subjects attending metabolic clinic who were suggested to use long term sensor due to persistent hyperglycemia and hypoglycemia
  Interventions: Device: Long term sensor

INTERVENTIONS:
Device: Long term sensor — Observational study including subjects using long term sensor according to local guidelines and patients preferences

SUMMARY:
The implantable Eversense ® CGM System obtained CE marking in 2016 for the 90-day device and in 2017 for the 180-day device.There is interest in real-world clinical evidence on the use of Eversense regarding changes in HbA1c and time in range (TIR), time below range (TBR), and time above range (TAR) in patients with type 1 diabetes. This is a prospective, multi-center, observational clinical study among adult participants aged 18 years or older with T1D and Eversense CGM System-naïve aimed to evaluate the change in HbA1c and glucometric parameters (TIR, TAR, TBR, mean daily glucose and standard deviation) in patients with T1D from multiple clinics in Italy using the Eversense CGM System for a 6-month time period.

DETAILED DESCRIPTION:
A new continuous glucose monitoring system (CGM), the Eversense ® CGM System (Company Senseonics, Inc., location of Company Germantown, MD) has been developed and commercially introduced in the last 3 years. This system may overcome drawbacks and limitations of traditional transcutaneous CGM systems. It consists of a fully implantable sensor lasting up to 180 days, a removable smart transmitter providing unique on-body vibratory alerts, and a mobile medical app (MMA) displaying glucose information captured and calculated by the transmitter. The app generates pop-up messages and alerts for glucose values crossing low and high thresholds, rate of change of glucose exceeding pre-set limits, and predicted low and high glucose levels. Glucose data are uploaded and stored in the cloud. Data from the cloud can be analyzed to provide different glucometric parameters such as time in range (TIR, 70-180 mg/dL), time below range (TBR, <70mg/dL), time above range (TAR, >180 mg/dL), mean daily glucose levels, and standard deviation (SD). The safety and accuracy of the new system has been evaluated in the PRECISE, PRECISE II and the PRECISION studies. The accuracy of the system is very high and no serious adverse events and very few adverse events have been reported in pivotal trials. Among adverse events, redness/erythema, bruising and pain at the sensor insertion site occurred. The purpose of this analysis will be to evaluate the change in HbA1c and in glucometric parameters, such as TIR, TBR, TAR, mean daily glucose, and SD in patients with T1D from multiple clinics in Italy using the Eversense CGM System for a 6-month time period. This is a prospective, multi-center, observational clinical research study among adult participants aged 18 years or older with T1D across several diabetes-care centers in Italy. Patients will be required to be Eversense CGM System-naïve. Patients will be trained on the Eversense CGM System use before sensor insertion, as suggested by the current clinical practice recommendations. Specifically, they will be instructed about the principles of the sensor technology, the operational aspects of the device, and the interpretation of displayed data. No specific therapeutic recommendations will be suggested to adjust pre-meal insulin dosing. Patients will be advised to take an action when alerts will be asserted, according to general recommendations, including checking the glucose value using a traditional blood glucose meter. The following parameters will be collected for each patient: HbA1c (measured using high-performance liquid chromatography) within two months before sensor implantation and 6 months after the implantation, disease duration, prior use of CGM, and insulin therapy delivery mode (MDI or CSII). The Eversense CGM System consists of an implantable, fluorescence-based, long-term sensor; the smart transmitter worn on top of the skin above the sensor; and the medical mobile app (MMA) which operates on a mobile device (smart phone, smart watch, or iPad) and provides real-time monitoring of current and historical glucose values. The long-term sensor will be implanted by trained endocrinologists into the subcutaneous tissue of the upper arm at the end of the deltoid muscle in all patients. Patients will be registered in the Eversense Data Management System (DMS) allowing automatic uploading of sensor glucose data. Study participants will be followed according to local practice. The euglycemic target (TIR, glucose 70-180 mg/dL), TAR (glucose >180 mg/dL), TBR (glucose <70 mg/dL), mean overall daily glucose, and mean SD, will be collected from the DMS over the first 2 weeks after the first sensor implantation (baseline) and 2 weeks before the 6-month visit. HbA1c and CGM metric changes in patients using CSII and MDI treatment for insulin delivery, and in patients who were CGM-naïve and prior CGM users will be assessed to observe the differences by prior CGM use and method of insulin delivery. Specifically, patients will be categorized into four different subgroups: CSII and prior CGM use, CSII and CGM naïve, MDI and prior CGM use, and MDI and CGM naïve. Appropriate tests will be performed using SPSS (Statistical Package for Social Science) 23 for Macintosh. Variables not normally distributed will be analyzed with non parametric test or if necessary a 2-step rank transformation will be applied to normalize the variables. All patients will be informed about the finality of the research and they will be required to give informed consent in order to analyze data collected by the DMS. They will receive all scheduled visits according to clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes
* Age >18 years
* Eversense ® CGM System-naïve

Exclusion Criteria:

* candidates for a MRI during sensor wear
* critically ill including hospitalization
* known contradiction to dexamethasone
* required intravenous mannitol or mannitol irrigation solutions
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants aged 18 years or older who were suggested to wear long term sensor.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-06-05 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
HbA1c (%) | six months
  Measured by High Performance Liquid Chromatography
Time in Range (%) | six months
  Collection from diabetes management system
Time Below Range (%) | six months
  Collection from diabetes management system
Time Above Range (%) | six months
  Collection from diabetes management system
Mean Daily Glucose (mmol/l) | six months
  Collection from diabetes management system
Glucose Standard Deviation (mmol/L) | six months
  Collection from diabetes management system

CONTACTS AND LOCATIONS:
Locations (1):
- University Magna Graecia, Catanzaro, Italy

REFERENCES:
- [Derived] Irace C, Cutruzzola A, Nuzzi A, Assaloni R, Brunato B, Pitocco D, Tartaglione L, Di Molfetta S, Cignarelli A, Laviola L, Citro G, Lovati E, Gnasso A, Tweden KS, Kaufman FR. Clinical use of a 180-day implantable glucose sensor improves glycated haemoglobin and time in range in patients with type 1 diabetes. Diabetes Obes Metab. 2020 Jul;22(7):1056-1061. doi: 10.1111/dom.13993. Epub 2020 Feb 27. PMID 32037699